CLINICAL TRIAL: NCT04801459
Title: A Single Center Randomized Prospective Study on the Peristaltic Direction of Gastrointestinal Anastomosis in Roux-en-Y Reconstruction After Distal Curative Gastrectomy for Gastric Cancer
Brief Title: Study on the Peristaltic Direction of GI Anastomosis in Roux-en-Y Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DJY002
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Peristaltic Direction; Roux-en-Y Gastrointestinal Anastomosis; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiperistaltic direction of gastrointestinal anastomosis in Roux-en-Y reconstruction group (Experimental): The isoperistaltic anastomosis represents the peristalsis direction of remnant stomach and jejunal efferent loop was consistent.
  Interventions: Procedure: Direction procedure of gastrointestinal anastomosis in Roux-en-Y reconstruction
- Isoperistaltic direction of gastrointestinal anastomosis in Roux-en-Y reconstruction group (Active Comparator): The antiperistaltic anastomosis represents the peristalsis direction of remnant stomach and jejunal efferent loop was opposite.
  Interventions: Procedure: Direction procedure of gastrointestinal anastomosis in Roux-en-Y reconstruction

INTERVENTIONS:
Procedure: Direction procedure of gastrointestinal anastomosis in Roux-en-Y reconstruction — In this study, intervention methods include two kind directions of gastrointestinal anastomosis in Roux-en-Y reconstruction after distal curative gastrectomy for gastric cancer. One is the isoperistaltic anastomosis, representing the peristalsis direction of remnant stomach and jejunal efferent loop was consistent. The other is the antiperistaltic anastomosis, representing the peristalsis direction of remnant stomach and jejunal efferent loop was opposite.

SUMMARY:
The aim of this study is intending to provide the optimal procedures of the peristaltic direction of gastrointestinal anastomosis in Roux-en-Y reconstruction after distal curative gastrectomy for gastric cancer, which can provide the best operation mode of Roux-en-Y anastomosis in digestive tract reconstruction during distal gastrectomy for reducing postoperative complications and improving quality of life for patients.

DETAILED DESCRIPTION:
In this study, all 148 the included patients will underwent the distal curative gastrectomy for gastric cancer and will be performed the Roux-en-Y reconstruction for gastrointestinal anastomosis. Of them, 74 patients will be randomized in the group undergoing with the isoperistaltic anastomosis in the Roux-en-Y reconstruction procedure. Meanwhile, the other 74 cases will be randomized in the group undergoing with the antiperistaltic anastomosis in the Roux-en-Y reconstruction procedure. Then, we will evaluate the differencies of effects of early recovery postoperatively (exhaust, defecation, eating, residual stomach peristalsis, length of hospital stay, etc.) and late gastrointestinal effects (bile reflux, residual gastritis, gastric emptying function, etc.) between above two group of patients, which will make an important contribution to reduce medical costs and potential improvements of the prognosis after distal curative gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) Pathological examination confirmation the adenocarcinoma of stomach before surgery
* 2) Physical conditions compliance with the requirements for curative gastrectomy
* 3) Consent to undergo the D2 lymphadenectomy, and the dissected proportion of stomach no less than 2/3
* 4) Comply with the protocol during the whole study period
* 5) No neoadjuvant therapy administration
* 6) Sign informed consent and permission of withdraw in the whole study period
* 7) Consent to provide the tissue specimens after surgery for this study
* 8) Estimation the overall survival after surgery no less than 6 months
* 9) No anesthesia or operation contraindication disease
* 10) cT1-4N0-2M0 stage demonstration by CT and endoscopic ultrasonography examinations
* 11) Negative cytological detection in operation
* 12) No seriously concomitance's diseases
* 13) Karnofsky Performance Scores (KPS) more than 60
* 14) Examined lymph node count no less than 16

Exclusion Criteria:

* 1) Women during pregnant stage and breast-feed stage
* 2) Women of childbearing age without any contraceptive measures
* 3) Severe congestive heart failure, frequent arrhythmia, or myocardial infarction within 12 months
* 4) Immunosuppressive therapists for organ transplantation
* 5) Seriously uncontrolled recurrent infection
* 6) other malignant tumors
* 7) No abilities of self-knowledge or mental disorders
* 8) Participating in other clinical trials
* 9) Siewert I and II esophagogastric junction tumors
* 10) Serious internal diseases obstruction surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Early postoperative recovery results | Within 1 month after surgery
  Differences of effects of early recovery postoperatively (exhaust, defecation, eating, residual stomach peristalsis, length of hospital stay, etc.)
Late postoperative recovery results | 1 year after surgery
  Differences of late gastrointestinal effects (bile reflux, residual gastritis, gastric emptying function, etc.)

OTHER OUTCOMES:
Postoperative complications | Within 1 month after surgery
  Postoperative incision infection, anastomotic leakage, intestinal obstruction, reoperation and readmission, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04801459/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04801459/SAP_001.pdf
  • Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04801459/ICF_002.pdf